CLINICAL TRIAL: NCT06207370
Title: A Double-blind Placebo-controlled Study to Assess the Safety and Efficacy of Oral Tafenoquine Plus Standard of Care Versus Placebo Plus Standard of Care in Patients Hospitalized for Babesiosis
Brief Title: Oral Tafenoquine Plus Standard of Care Versus Placebo Plus Standard of Care for Babesiosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: 60 Degrees Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQ-BA-2024-1
Record Dates: First submitted 2023-12-21; First posted 2024-01-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Babesiosis
Keywords: babesiosis
MeSH Terms: conditions — Babesiosis | interventions — tafenoquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): TQ: 2 x 100 mg TQ tablets orally on Days 1, 2, 3, and 4
  Interventions: Drug: Tafenoquine
- Group 2 (Placebo Comparator): Placebo: 2 x 100 mg placebo tablets orally on Days 1, 2, 3, and 4
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tafenoquine — Oral Tafenoquine
  Arms: Group 1
Other: Placebo — Placebo
  Arms: Group 2

SUMMARY:
This study is a double-blind, randomized, multisite, placebo-controlled trial comparing the safety and efficacy of TQ versus placebo in patients hospitalized for babesiosis with low risk for relapsing disease who will also be administered a standard-of-care antimicrobial regimen (A/A) that is recommended in the 2020 IDSA guideline on the diagnosis and management of babesiosis.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, multisite, placebo-controlled trial comparing the safety and efficacy of TQ versus placebo in patients hospitalized for babesiosis with low risk for relapsing disease who will also be administered a standard-of-care antimicrobial regimen (A/A) that is recommended in the 2020 IDSA guideline on the diagnosis and management of babesiosis.

Patients hospitalized for a diagnosis of babesiosis, who have received A/A for <48 hours (h) prior to randomization or are about to receive A/A, will be asked to provide written informed consent and will undergo eligibility screening including medical history, physical examination, prior and concomitant medications, blood chemistry and hematology, glucose-6-phosphate dehydrogenase (G6PD) deficiency testing, blood smear for diagnostic confirmation of babesiosis, pregnancy testing for females of child-bearing potential, and assessment of risk factors for relapsing babesiosis. The screening period will last a maximum of two days. The first day of dosing with TQ or placebo will be Day 1 and will be done while the patient is still hospitalized.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 years.
* Laboratory confirmed infection with Babesia.
* Exhibiting at least one self-reported clinical symptoms of babesiosis.
* Able and willing to give written informed consent.
* Expected to be hospitalized at the time of or following informed consent and still hospitalized on the day of randomization and start of investigational products.
* Willing to complete the study activities and assessments.
* Must agree not to enroll in another study of an investigational agent prior to completion of the study.
* Able to take oral medications.
* If female of reproductive age, must agree to use an acceptable method of birth control.
* Adequate venous access.
* Blood hemoglobin ≥ 7 g/dL.

Exclusion Criteria:

* Have any contraindications to TQ.
* Have any contraindication for azithromycin or atovaquone.
* Any concomitant significant illness unrelated to babesiosis.
* Receipt of any experimental treatment for babesiosis.
* Taking any excluded concomitant medication.
* Current or planned treatment with quinine while participating in the study.
* Positive pregnancy test.
* If A/A was initiated more than 48h prior to randomization and parasitemia is not >1%.
* Azithromycin or atovaquone administered in the last 12 months to treat babesiosis, and, in the opinion of the investigator, high likelihood that current infection represents a relapse or continuation of disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Time to sustained clinical resolution | Day 1 to 90
  Time to sustained clinical resolution of all the following symptoms of babesiosis: sweats, joint aches, cough, loss of appetite, muscle aches, headache, chills or shivering, feeling hot or feverish, nausea, fatigue (low energy or tiredness), and vomiting. The time to achieve sustained clinical resolution will be the date when patients first self-report a 7-day period without these symptoms relative to the start of tafenoquine or placebo treatment.

SECONDARY OUTCOMES:
Difference in TTMC between TQ and placebo | Day 1 to 90
  Difference in TTMC between TQ and placebo from Day 1 to Day 90 (± 7 days). Molecular cure is defined as the time to the first instance of a negative NAT.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No